CLINICAL TRIAL: NCT01298661
Title: Evaluation of Reliability, Sensitivity and Validity of the Six Minute Step Test in Patients With Chronic Obstructive Pulmonary Disease and Its Relation With Predictors Markers of Risk of Death
Brief Title: Reliability, Sensitivity and Validity of the 6 Minute Step Test in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Valeria Amorim Pires Di Lorenzo, PhD, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TD6reprod
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exercise Test; Reproducibility of Results; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy Young Subjects (Other): Subjects apparently healthy, with age of 18 to 27 years old.
  Interventions: Other: Six-minute Step Test
- Healthy Elderly subjects (Other): Subjects apparently healthy, with age of 60 to 75 years old.
  Interventions: Other: Six-minute Step Test
- COPD Patients (Other): Patients with clinical and spirometric diagnosis of COPD
  Interventions: Other: Six-minute Step Test

INTERVENTIONS:
Other: Six-minute Step Test — The patients underwent a test where they need to step up and down a 20cm test during six minutes.
  Other Names: Exercise Test

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) leads to a reduction in exercise capacity that affects the quality of life and increases mortality of these patients. So, exercise tests are considered as an essential component of the clinical evaluation of the patients with COPD. The objective of this study is to evaluate the reproducibility sensitivity and validity of the Six Minute Step Test (6MST) in patients with COPD and in health volunteers, and verify its relation with the "Body-Mass Index, Airways Obstruction, Dyspnea and Exercise Capacity" Index (BODE). This Observational, Transversal, Prospective study will be conducted in the "Special Unit of Respiratory Physiotherapy", of the "Federal University of São Carlos". To participate in this study, 120 subjects, both gender, will be invited and will be allocated in five groups: Group I (30 healthy young subjects of 17 to 27 years old), Group II (30 healthy elderly individuals of 60 to 75 years old), and patients COPD, 60 to 80 years old, with mild, moderate, severe and very severe obstruction determined by the forced expiratory volume in one second (FEV1) by forced vital capacity (FVC) relation "FEV1/FVC" <70% and FEV1 in predict percentage < 80% composing the Group III (20 COPD patients in GOLD stage I), Group IV (20 COPD patients in GOLD stage II) and Group V (20 patients COPD stages III and IV). All subjects will be submitted to body composition and anthropometric assessment, pulmonary function test, three 6-minutes walk test (6MWT) and three 6MST. Furthermore, the patients of the groups III, IV and V will answer the Modified Medical Research Council (mMRC) scale, and BODE index will be calculated to each of them.

ELIGIBILITY:
Inclusion Criteria:

* Young and elderly healthy subjects presented pulmonary function within the normal range, confirmed by spirometry
* Patients with clinical and spirometric diagnosis of COPD

Exclusion Criteria:

* Lung disease exacerbated
* Decompensated heart disease
* Rheumatic, neurological or orthopedic disease, preventing them from doing the tests by limiting the exercise
* Peripheral oxygen saturation < 80% without physical effort
* Subjects who does not complete the first day of evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Amorim Pires Di Lorenzo, PhD, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Unidade Especial de Fisioterapia Respiratória, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Baarends EM, Schols AM, Mostert R, Wouters EF. Peak exercise response in relation to tissue depletion in patients with chronic obstructive pulmonary disease. Eur Respir J. 1997 Dec;10(12):2807-13. doi: 10.1183/09031936.97.10122807. PMID 9493665
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Cahalin LP, Mathier MA, Semigran MJ, Dec GW, DiSalvo TG. The six-minute walk test predicts peak oxygen uptake and survival in patients with advanced heart failure. Chest. 1996 Aug;110(2):325-32. doi: 10.1378/chest.110.2.325. PMID 8697828
- [Background] Cataneo DC, Cataneo AJ. Accuracy of the stair climbing test using maximal oxygen uptake as the gold standard. J Bras Pneumol. 2007 Mar-Apr;33(2):128-33. doi: 10.1590/s1806-37132007000200005. English, Portuguese. PMID 17724530
- [Background] Casanova C, Cote C, Marin JM, Pinto-Plata V, de Torres JP, Aguirre-Jaime A, Vassaux C, Celli BR. Distance and oxygen desaturation during the 6-min walk test as predictors of long-term mortality in patients with COPD. Chest. 2008 Oct;134(4):746-752. doi: 10.1378/chest.08-0520. Epub 2008 Jul 14. PMID 18625667
- [Background] Casas A, Vilaro J, Rabinovich R, Mayer A, Barbera JA, Rodriguez-Roisin R, Roca J. Encouraged 6-min walking test indicates maximum sustainable exercise in COPD patients. Chest. 2005 Jul;128(1):55-61. doi: 10.1378/chest.128.1.55. PMID 16002916
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Dal Corso S, Duarte SR, Neder JA, Malaguti C, de Fuccio MB, de Castro Pereira CA, Nery LE. A step test to assess exercise-related oxygen desaturation in interstitial lung disease. Eur Respir J. 2007 Feb;29(2):330-6. doi: 10.1183/09031936.00094006. Epub 2006 Oct 18. PMID 17050559
- [Background] Dourado VZ, Tanni SE, Vale SA, Faganello MM, Sanchez FF, Godoy I. Systemic manifestations in chronic obstructive pulmonary disease. J Bras Pneumol. 2006 Mar-Apr;32(2):161-71. doi: 10.1590/s1806-37132006000200012. English, Portuguese. PMID 17273586
- [Background] Dourado VZ, Antunes LC, Tanni SE, de Paiva SA, Padovani CR, Godoy I. Relationship of upper-limb and thoracic muscle strength to 6-min walk distance in COPD patients. Chest. 2006 Mar;129(3):551-7. doi: 10.1378/chest.129.3.551. PMID 16537851
- [Background] Enright PL, McBurnie MA, Bittner V, Tracy RP, McNamara R, Arnold A, Newman AB; Cardiovascular Health Study. The 6-min walk test: a quick measure of functional status in elderly adults. Chest. 2003 Feb;123(2):387-98. doi: 10.1378/chest.123.2.387. PMID 12576356
- [Background] Fromer L, Cooper CB. A review of the GOLD guidelines for the diagnosis and treatment of patients with COPD. Int J Clin Pract. 2008 Aug;62(8):1219-36. doi: 10.1111/j.1742-1241.2008.01807.x. Epub 2008 Jun 28. PMID 18547365
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Soler-Cataluna JJ, Sanchez-Sanchez L, Martinez-Garcia MA, Sanchez PR, Salcedo E, Navarro M. Mid-arm muscle area is a better predictor of mortality than body mass index in COPD. Chest. 2005 Oct;128(4):2108-15. doi: 10.1378/chest.128.4.2108. PMID 16236862
- [Background] Pitta F, Troosters T, Spruit MA, Probst VS, Decramer M, Gosselink R. Characteristics of physical activities in daily life in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 May 1;171(9):972-7. doi: 10.1164/rccm.200407-855OC. Epub 2005 Jan 21. PMID 15665324
- [Background] Pinto-Plata VM, Cote C, Cabral H, Taylor J, Celli BR. The 6-min walk distance: change over time and value as a predictor of survival in severe COPD. Eur Respir J. 2004 Jan;23(1):28-33. doi: 10.1183/09031936.03.00034603. PMID 14738227
- [Background] Mahler DA, Wells CK. Evaluation of clinical methods for rating dyspnea. Chest. 1988 Mar;93(3):580-6. doi: 10.1378/chest.93.3.580. PMID 3342669
- [Background] Leung AS, Chan KK, Sykes K, Chan KS. Reliability, validity, and responsiveness of a 2-min walk test to assess exercise capacity of COPD patients. Chest. 2006 Jul;130(1):119-25. doi: 10.1378/chest.130.1.119. PMID 16840391
- [Background] Hadeli KO, Siegel EM, Sherrill DL, Beck KC, Enright PL. Predictors of oxygen desaturation during submaximal exercise in 8,000 patients. Chest. 2001 Jul;120(1):88-92. doi: 10.1378/chest.120.1.88. PMID 11451821
- [Background] Kovelis D, Segretti NO, Probst VS, Lareau SC, Brunetto AF, Pitta F. Validation of the Modified Pulmonary Functional Status and Dyspnea Questionnaire and the Medical Research Council scale for use in Brazilian patients with chronic obstructive pulmonary disease. J Bras Pneumol. 2008 Dec;34(12):1008-18. doi: 10.1590/s1806-37132008001200005. English, Portuguese. PMID 19180335
- [Background] Knudson RJ, Lebowitz MD, Holberg CJ, Burrows B. Changes in the normal maximal expiratory flow-volume curve with growth and aging. Am Rev Respir Dis. 1983 Jun;127(6):725-34. doi: 10.1164/arrd.1983.127.6.725. PMID 6859656
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Derived] Pessoa BV, Arcuri JF, Labadessa IG, Costa JN, Sentanin AC, Di Lorenzo VA. Validity of the six-minute step test of free cadence in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2014 May-Jun;18(3):228-36. doi: 10.1590/bjpt-rbf.2014.0041. PMID 25003275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment occurred from February 2011 until July 2012. The COPD patients were those referred to pulmonary rehabilitation on Unidade Especial de Fisioterapia Respiratória and the health individuals were recruited by invitation using posters on the University region.
Period: Overall Study
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Started | 33 | 24 | 34
Completed | 31 | 24 | 32
Not Completed | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: In the group of health young subjects there were a loss of 2 individuals who did not completed the evaluations.
  In the group of COPD patients there was a loss of 2 patients who did not completed the evaluations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients | Total
Number analyzed (Participants) | 31 | 24 | 32 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 6 | 9 | 46
  >=65 years | 0 | 18 | 23 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 22.7 (2.52) | 68.9 (6.75) | 68.6 (10.3) | 52.3 (23.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 8 | 35
  Male | 16 | 12 | 24 | 52
Region of Enrollment [Number; unit: participants]
  Brazil | 31 | 24 | 32 | 87

OUTCOME MEASURES:

1. Primary Outcome: First "Six Minute Step Test" Performance
Description: This test will be conducted by the "Rater 1", the patient will step up and down a 20cm step during six minute. The performance will be evaluated by the number of the steps.
Time Frame: First day or second day of the protocol (random)
Population: 2 COPD patients and 2 healthy young individuals were excluded since they did not appeared in the second day of evaluation.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
steps | 166.4 (36.4) | 114.0 (29.2) | 76.6 (19.6)

2. Primary Outcome: Second "Six Minute Step Test" Performance
Description: This test will be conducted by the "Rater 1", the patient will step up and down a 20cm step during six minutes. The performance will be evaluated by the number of the climbs.
Time Frame: On the first or second day of evaluation (random), 30 minutes after the first 6MST.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
steps | 170.7 (40.6) | 114.5 (33.5) | 82.4 (20.7)

3. Primary Outcome: Third "Six Minute Step Test" Performance
Description: This test will be conducted by the "Rater 2", the patient will step up and down a 20cm step during six minutes. The performance will be evaluated by the number of the climbs.
Time Frame: On the third day of evaluation, seven days after the first day of evaluation. Since it was performed in the same day of the third 6MWT, the choice of the first test was random, and there was a 30 minute interval between them.
Population: 2 COPD patients and 2 healthy young individuals were excluded from the study since they did not appeared in the second day of evaluation. 3 COPD patient Analysis Population Description: s and 5 elderly subjects didn't show on the third day of evaluation, then, they were just excluded in the analysis of the variables collected in this day.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
steps | 172.3 (36.3) | 111.3 (32.9) | 86.4 (22.0)

4. Secondary Outcome: First "Six Minute Walk Test" Distance
Description: This test will be conducted by the "Rater 1", the subject will walk as far as it can in a 30m corridor during 6 minutes. The performance will be the distance (meters)that it walk.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
meter | 643.5 (63.1) | 504.5 (119) | 380.4 (107.8)

5. Secondary Outcome: Second "Six Minute Walk Test" Distance
Description: as for outcome 4
Time Frame: On the first or second day of evaluation (random), 30 minutes after the first 6MWT.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
meter | 648.2 (81.9) | 513.6 (84.3) | 391.0 (94.0)

6. Secondary Outcome: Third "Six Minute Walk Test" Distance
Description: This test will be conducted by the "Rater 2", the subject will walk as far as it can in a 30m corridor during 6 minutes. The performance will be the distance (meters)that it walk.
Time Frame: On the third day of evaluation, seven days after the first day of evaluation. Since it was performed in the same day of the third 6MST, the choice of the first test was random, and there was a 30 minute interval between them.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
meter | 648.3 (73.9) | 502 (112.4) | 392.4 (93.0)

7. Secondary Outcome: "Body-Mass Index, Airflow Obstruction, Dyspnea, Exercise Capacity" Index (BODE Index)
Description: It was evaluated only in the COPD patients. BODE index is a prognostic index used in COPD patients, it is a 0-10 scale, where lower values means better prognostic. It is composed by other commonly used evaluations tools in COPD, Forced Expiratory Volume in the First second (from spirometry); classification in the scale ranging from 0-3, Body-mass index, classification in the scale ranging from 0-1; Six-minute walk test distance, classification in the scale ranging from 0-3 and referred dyspnea, classification in the scale ranging from 0-3.
  It was only used the total score (0-10)
Time Frame: Second day
Population: 2 COPD were excluded since they did not appeared in the second day of evaluation. The other two populations were not verified, since the measure is specific for COPD patients
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- COPD Patients: Patients with clinical and spirometrical diagnosis of Chronic Obstructive Pulmonary Disease
Arm/Group | COPD Patients
Number analyzed (Participants) | 32
units on a scale | 3 [1 to 4]

8. Secondary Outcome: First "Six Minute Walk Test" Exertion Perception
Description: This test was conducted by the "Rater 1", the subject walked as far as it could in a 30m corridor during 6 minutes. The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
units on a scale | 1 [0 to 5] | 0.5 [0 to 5] | 1 [0 to 5]

9. Secondary Outcome: Second "Six Minute Walk Test" Exertion Perception
Description: This test will be conducted by the "Rater 1", the subject will walk as far as it can in a 30m corridor during 6 minutes. The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: First day or second day of the protocol (random), 30 minutes after the first 6MWT
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
units on a scale | 0.5 [0 to 5] | 0.5 [0 to 6] | 1 [0 to 4]

10. Secondary Outcome: Third "Six Minute Walk Test" Exertion Perception
Description: This test will be conducted by the "Rater 2", the subject will walk as far as it can in a 30m corridor during 6 minutes. The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
units on a scale | 1 [0 to 3] | 1 [0 to 5] | 2 [0 to 5]

11. Secondary Outcome: First "Six Minute Step Test" Exertion Perception
Description: This test will be conducted by the "Rater 1", the patient will step up and down one 20cm step during six minute. The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
units on a scale | 2 [0 to 5] | 2.5 [0 to 7] | 2 [0 to 7]

12. Secondary Outcome: Second "Six Minute Step Test" Exertion Perception
Description: This test will be conducted by the "Rater 1", the patient will step up and down one 20cm step during six minute.The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: First day or second day of the protocol (random), 30 minutes after the first 6MST
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
units on a scale | 2 [0 to 7] | 1.5 [0 to 6] | 2.5 [0 to 7]

13. Secondary Outcome: Third "Six Minute Step Test" Exertion Perception
Description: This test will be conducted by the "Rater 2", the patient will step up down one 20cm step during six minute. The Exertion Perception will be evaluated using BORG scale. This scale is a self-reported scale, which range from 0 to 10, where 0 means none exertion perception and 10 means very intense exertion perception (the highest the patient has ever felt). Lower values means that the patient feel less discomfort.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
units on a scale | 1 [0 to 6] | 2 [0 to 7] | 2.5 [0 to 8]

14. Secondary Outcome: First "Six Minute Walk Test" Peripheral Oxygen Saturation
Description: This test will be conducted by the "Rater 1", the subject will walk as far as it can in a 30m corridor during 6 minutes. It will be evaluated by a pulse oxymeter.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
% of hemoglobin | 96.7 (1.3) | 94.5 (1.7) | 90.4 (3.15)

15. Secondary Outcome: Second "Six Minute Walk Test" Peripheral Oxygen Saturation
Description: as for outcome 14
Time Frame: ,First day or second day of the protocol (random) 30 minutes after the first 6MWT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
% of hemoglobin | 96.4 (1.81) | 95.1 (1.48) | 90.3 (3.33)

16. Secondary Outcome: Third "Six Minute Walk Test" Peripheral Oxygen Saturation
Description: This test will be conducted by the "Rater 2", the subject will walk as far as it can in a 30m corridor during 6 minutes. It will be evaluated by a pulse oxymeter.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
% of hemoglobin | 96.1 (1.6) | 94.7 (2.0) | 89.7 (3.3)

17. Secondary Outcome: First "Six Minute Step Test" Peripheral Oxygen Saturation
Description: This test will be conducted by the "Rater 1", the patient will step up and down one 20cm step during six minute. It will be evaluated by a pulse oxymeter.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
% of hemoglobin | 95.8 (1.3) | 95 (1.9) | 90.1 (3.9)

18. Secondary Outcome: Second "Six Minute Step Test" Peripheral Oxygen Saturation
Description: This test will be conducted by the "Rater 1", the patient will step up and down one 20cm step during six minute. It will be evaluated by a pulse oxymeter .
Time Frame: First day or second day of the protocol (random) ,30 minutes after the first 6MST
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
% of hemoglobin | 96 (1.6) | 94.9 (1.8) | 90.5 (2.8)

19. Secondary Outcome: Third "Six Minute Step Test" Peripheral Oxygen Saturation
Description: This test will be conducted by the "Rater 2", the patient will step up and down one 20cm step during six minute. It will be evaluated by a pulse oxymeter.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: % of hemoglobin
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
% of hemoglobin | 95.8 (1.3) | 94.9 (1.8) | 90.3 (3.1)

20. Secondary Outcome: First "Six Minute Walk Test" Heart Rate
Description: This test will be conducted by the "Rater 1", the subject will walk as far as it can in a 30m corridor during 6 minutes. It will be evaluated by a cardio monitor.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
bpm | 143 (15) | 115 (11) | 113 (11)

21. Secondary Outcome: Second "Six Minute Walk Test" Heart Rate
Description: This test will be conducted by the "Rater 1", the subject will walk as far as it can in a 30m corridor during 6 minutes. It will be evaluated by a cardio monitor at rest and every two minutes of the test.
Time Frame: First day or second day of the protocol (random), 30 minutes after the first 6MWT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
bpm | 144 (13) | 115 (9) | 112 (11)

22. Secondary Outcome: Third "Six Minute Walk Test" Heart Rate
Description: This test will be conducted by the "Rater 2", the subject will walk as far as it can in a 30m corridor during 6 minutes. It will be evaluated by a cardio monitor.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
bpm | 145 (10) | 112 (13) | 114 (13)

23. Secondary Outcome: First "Six Minute Step Test" Heart Rate
Description: This test will be conducted by the "Rater 1", the patient will step up and down a 20cm step during six minute. It will be evaluated by a cardio monitor.
Time Frame: First day or second day of the protocol (random)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
bpm | 154 (11) | 116 (11) | 117 (10)

24. Secondary Outcome: Second "Six Minute Step Test" Heart Rate
Description: as for outcome 23
Time Frame: First day or second day of the protocol (random), 30 minutes after the first 6MST
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 24 | 32
bpm | 159 (6.7) | 118 (8.7) | 117 (12)

25. Secondary Outcome: Third "Six Minute Step Test" Heart Rate
Description: This test will be conducted by the "Rater 2", the patient will step up and down a 20cm step during six minute. It will be evaluated by a cardio monitor.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Number analyzed (Participants) | 31 | 19 | 29
bpm | 156 (11) | 117 (9.3) | 116 (15)

ADVERSE EVENTS:
Description: Adverse events were not assessed in this study.
Arm/Group | Healthy Young Subjects | Healthy Elderly Subjects | COPD Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The enrolled patient's and subject's numbers were smaller than the estimated for healthy elders and different COPD groups, because of the low acceptance of a three days evaluation protocol. So COPD patients were analyzed in a single group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No